CLINICAL TRIAL: NCT02820987
Title: Pharmacokinetics and Pharmacodynamic (PK/PD) of Extended-infusion Meropenem, Piperacillin-tazobactam and Cefepime in the Early Phase of Septic Shock
Brief Title: PK/PD of Extended-infusion Meropenem, Piperacillin-tazobactam and Cefepime in the Early Phase of Septic Shock
Acronym: PAACS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/493
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2018-07

CONDITIONS: Septic Shock
Keywords: Septic shock, Beta Lactams, Extended infusion, PK/PD
MeSH Terms: conditions — Shock, Septic | interventions — Meropenem; Piperacillin, Tazobactam Drug Combination; Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MEROPENEM (Active Comparator): After enrollment, patients of MEROPENEM arm will receive an initial 2g bolus of MEROPENEM and 2g infusion over 3 hours every eight hours, during 48 hours, without modification of rhythm and dose according to renal function.
  Interventions: Drug: MEROPENEM
- PIPERACILLIN-TAZOBACTAM (Active Comparator): After enrollment, patients of PIPERACILLIN - TAZOBACTAM arm will receive an initial 4g bolus of PIPERACILLIN - TAZOBACTAM and a 16g continuous infusion per day, during 48 hours, without modification of rhythm and dose according to renal function.
  Interventions: Drug: PIPERACILLIN-TAZOBACTAM
- CEFEPIME (Active Comparator): After enrollment, patients of CEFEPIME arm will receive an initial 2g bolus of CEFEPIME and a 6g continuous infusion per day, during 48 hours, without modification of rhythm and dose according to renal function.
  Interventions: Drug: CEFEPIME

INTERVENTIONS:
Drug: MEROPENEM — Administration of MEROPENEM according to a protocol of extended infusion defining dose and duration of infusion.
  Arms: MEROPENEM
Drug: PIPERACILLIN-TAZOBACTAM — Administration of PIPERACILLIN-TAZOBACTAM according to a protocol of continuous infusion defining dose and duration of infusion.
  Arms: PIPERACILLIN-TAZOBACTAM
Drug: CEFEPIME — Administration of CEFEPIME according to a protocol of continuous infusion defining dose and duration of infusion.
  Arms: CEFEPIME

SUMMARY:
This study evaluates PK/PD of an extended-infusion protocol of meropenem, piperacillin-tazobactam and cefepime, in the early phase of septic shock.

DETAILED DESCRIPTION:
Beta Lactams are the keystones of shock septic treatment. Early phase of septic shock is a period of disturbed pharmacokinetics, with augmented renal clearance and distribution volume of hydrophilic drugs as Beta Lactams. Consequently, early phase of septic shock is a period at risk of underdosing Beta Lactam, which could increase the risk of clinical failure an mortality.

Data are available concerning underdosing of MEROPENEM, PIPERACILLIN-TAZOBACTAM and CEFEPIME, when administered in bolus.

No data exist concerning the achievement of a target of 100% of the whole interval above 4 time the superior breakpoint of Pseudomonas Aeruginosa according to EUCAST (European Committee on Antimicrobial Susceptibility Testing), during the 48 first hours of treatment of septic shock, when Beta Lactam are administered in extended infusion.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* Meropenem, piperacillin-tazobactam or cefepime started after enrollment

Exclusion Criteria:

* Pregnancy
* Central nervous system infection
* Burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving the PK/PD target | First 48 hours
  Proportion of patients achieving the target of 100% of 48 first hours of treatment above 4 time the upper critical breakpoint for Pseudomonas Aeruginosa

SECONDARY OUTCOMES:
All cause mortality | 28th day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taccone FS, Laterre PF, Dugernier T, Spapen H, Delattre I, Wittebole X, De Backer D, Layeux B, Wallemacq P, Vincent JL, Jacobs F. Insufficient beta-lactam concentrations in the early phase of severe sepsis and septic shock. Crit Care. 2010;14(4):R126. doi: 10.1186/cc9091. Epub 2010 Jul 1. PMID 20594297
- [Derived] Winiszewski H, Despres C, Puyraveau M, Lagoutte-Renosi J, Montange D, Besch G, Floury SP, Chaignat C, Labro G, Vettoretti L, Clairet AL, Capellier G, Vivet B, Piton G. beta-lactam dosing at the early phase of sepsis: Performance of a pragmatic protocol for target concentration achievement in a prospective cohort study. J Crit Care. 2022 Feb;67:141-146. doi: 10.1016/j.jcrc.2021.10.023. Epub 2021 Nov 9. PMID 34768176